CLINICAL TRIAL: NCT01423994
Title: Syncope: Pacing or Recording in the Later Years (SPRITELY)
Brief Title: Syncope: Pacing or Recording in the Later Years
Acronym: Spritely
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Canadian Institutes of Health Research (CIHR) (Other Government)
Collaborators: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Dr. Bob Sheldon, Professor of Cardiac Sciences, Medicine and Medical Genetics, University of Calgary
Organization: University of Calgary (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIHR#230880
Record Dates: First submitted 2011-08-22; First posted 2011-08-26 (Estimated); Last update posted 2019-05-16 (Actual); Status verified 2019-05

CONDITIONS: Syncope; Heart Block; Conduction Disorder of the Heart
Keywords: syncope; fainting; implantable loop recorder; pacemaker; heart block; bifascicular heart block
MeSH Terms: conditions — Syncope; Heart Block; Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- implantable loop recorder (Active Comparator)
  Interventions: Procedure: implantable loop recorder
- pacemaker (Active Comparator)
  Interventions: Procedure: pacemaker

INTERVENTIONS:
Procedure: pacemaker — A single or dual chamber pacemaker will be implanted according to the manufacturer's instructions for use with standard techniques.
  Either a single or dual chamber pacemaker will be permitted according to local practice unless the patient is in chronic or persistent atrial fibrillation, in which case a single chamber pacemaker will be used. The pacemaker configuration will be at the discretion of the investigator.
  Single chamber ventricular pacemakers will be programmed to activity responsiveness off in VVI mode, rates 50-120 bpm.
  Dual chamber pacemaker programming will be to DDD mode (50-120) with mode switch on.
  Arms: pacemaker
Procedure: implantable loop recorder — The implantable loop recorder will be programmed for automatic detection using settings of Low Heart Rate <50 bpm, High Heart Rate >165 bpm, and Pause > 3 seconds.
  Arms: implantable loop recorder

SUMMARY:
Syncope affects about 50% of Canadians, is the cause of 1 - 2% of all emergency room visits, and probably is responsible for CDN $250 million in health care spending each year. It is associated with decreased quality of life, trauma, loss of employment, and limitations in daily activities. It is a particular problem for older people, partly because of increased frailty, and partly because of a difficult differential diagnosis. One of the causes in older adults is intermittent complete heart block in the setting of bifascicular heart block, but they may also faint due to a variety of tachyarrhythmias, sick sinus syndrome, and several neurally mediated syncopes. Often treatment decisions should be made before the true cause is apparent.

DETAILED DESCRIPTION:
There are two general approaches to the patient with syncope and bifascicular block, a common substrate for intermittent heart block. The first is to assume that intermittent heart block is the cause, and simply implant a pacemaker. The second is to implant a digital ECG loop recorder with a lifespan of 2 - 3 years, determine the rhythm abnormalities during the next faint, and treat accordingly. Both approaches expose patients to a risk of fainting and its sequelae, and both carry device-related complications.Which approach is superior is unknown.

ELIGIBILITY:
Inclusion Criteria:

-Patients are eligible if they have:

* >1 syncopal spell within 1 year preceding enrollment, and
* bifascicular block on a 12-lead ECG, and
* Age > 50 years and
* written informed consent. Syncope will be defined based on history using a standardized form.

Exclusion Criteria:

-Patients will be excluded if they have criteria related to study strategies, including:

1. previous pacemaker, ICD, or Implantable Loop Recorder in situ,
2. ACC/AHA/HRS Class I indication for permanent pacing or ICD implantation,
3. left ventricular ejection fraction < 35% mandating ICD therapy,
4. contra-indication to a transvenous pacemaker such as artificial tricuspid valve or active sepsis.

   -Patients will also be excluded if a potential competing cause of syncope poses a threat to life, such as:
5. hypertrophic cardiomyopathy,
6. documented sustained ventricular tachycardia or
7. inducible, sustained monomorphic ventricular tachycardia on EP study.

   -They will be excluded if they have:
8. a history of myocardial infarction within 3 months prior to enrollment, and
9. a major chronic co-morbid medical condition that would preclude 24 months of follow-up.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2011-08; Primary Completion 2017-05 (Actual); Study Completion 2017-11-01 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure will be a composite of Major Adverse Study-Related Events (MASRE) in a 2-year observation period. | 2 years
  MASRE will capture the major consequences ensuing from both strategies, including 1) syncope, 2) symptomatic bradycardias, 3) asymptomatic complete heart block, 4) acute and chronic pacemaker and ILR complications, and 5) death.

SECONDARY OUTCOMES:
Secondary outcome measures will include total number of syncopal spells. | 2 years
Secondary outcome measures will include the likelihood of a first recurrence of syncope. | 2 years
Secondary outcome measures will include the physical trauma due to syncope. | 2 years
Secondary outcome measures will include quality of life of the participants. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Robert S Sheldon, MD, PhD, Principal Investigator — University of Calgary
Locations (17):
- Vanderbilt University, Nashville, Tennessee, United States
- Canada (11):
  - University of Calgary, Calgary, Alberta
  - Royal Alexandra Hospital, Edmonton, Alberta
  - Victoria Heart Institute, Victoria, British Columbia
  - St. Boniface Hospital, Winnipeg, Manitoba
  - Horizon Health Network New Brunswick, Saint John, New Brunswick
  - Mc Master University, Hamilton, Ontario
  - Queen's University, Kingston, Ontario
  - London Health Sciences Centre, London, Ontario
  - Montreal Heart Institute, Montreal, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec
  - Prairie Vascular Research Inc., Regina, Saskatchewan
- Japan (2):
  - University of Occupational and Environmental Health, Kitakyushu
  - Shwa General Hospital, Saitama
- University Malaya Medical Centre, Kuala Lumpur, Malaysia
- United Kingdom (2):
  - Kings College Hospital, London
  - James Cook University Hospital, Middlesbrough

REFERENCES:
- [Derived] Sheldon R, Talajic M, Tang A, Becker G, Essebag V, Sultan O, Baranchuk A, Ritchie D, Morillo C, Krahn A, Brignole M, Manns B, Maxey C, Raj SR; SPRITELY Investigators. Randomized Pragmatic Trial of Pacemaker Versus Implantable Cardiac Monitor in Syncope and Bifascicular Block. JACC Clin Electrophysiol. 2022 Feb;8(2):239-248. doi: 10.1016/j.jacep.2021.10.003. Epub 2021 Nov 24. PMID 35210082